CLINICAL TRIAL: NCT01048801
Title: Role and Effectiveness of Rapid Diagnostic Tests in Home-based Management of Malaria: Comparative Trials in Two Areas of High and Low Transmission in Uganda
Brief Title: Role and Effectiveness of Rapid Diagnostic Tests in Home-based Management of Malaria
Acronym: ACTUGA2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DBL -Institute for Health Research and Development (Other)
Collaborators: Ministry of Health, Uganda (Other Government); London School of Hygiene and Tropical Medicine (Other); Artemisinin-based Combination Therapy (Other)
Responsible Party: Principal Investigator, Pascal Magnussen, senior researcher, DBL -Institute for Health Research and Development
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTUGA2
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Fever; Malaria
Keywords: History of fever; measured fever
MeSH Terms: conditions — Fever; Malaria | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rapid diagnostic test and treatment (Active Comparator)
  Interventions: Device: Rapid diagnostic test
- Treatment without rapid daignostic test (Other)
  Interventions: Other: presumptive malaria treatment

INTERVENTIONS:
Device: Rapid diagnostic test — Use of rapid daignostic tests for diagnosis of malaria
  Arms: Rapid diagnostic test and treatment
Other: presumptive malaria treatment — Treatment of malariabased on clinical diagnosis without use of diagnostic test
  Arms: Treatment without rapid daignostic test

SUMMARY:
Most malaria deaths occur within 48 hours of onset of symptoms, and in rural areas with poor access to health facilities, home management of malaria (HMM) can improve the timeliness of treatment and reduce malaria mortality by up to 50%. In order to maximize both coverage and impact, ACTs should be deployed in HMM programmes, as well as in formal health facilities. Up to 80% of malaria cases are treated outside the formal health sector and shops are frequently visited as the first (and in some cases only) source of treatment. Strategies to deploy ACTs in Africa thus also need to examine the role of shops in home management and to ensure that drugs sold are appropriate. The current practice of presumptive treatment of any febrile illness as malaria (both at health facilities and in the context of HMM) based solely on clinical symptoms without routine laboratory confirmation, results in significant over-use of antimalarial drugs. With ACT being a more costly regimen, it is important to be more restrictive in its administration and rapid diagnostic tests (RDTs) provide a simple means of confirming malaria diagnosis in remote locations lacking electricity and qualified health staff.

This study therefore proposes to evaluate the feasibility, acceptability, and cost-effectiveness of using RDTs to improve malaria diagnosis and treatment by community-based drug distributors.The accuracy of RDTs, and the acceptability of this approach, will be evaluated in both low and high transmission areas.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 6 months and 5 years (< 5 years)reported with fever by the mother/ caretaker of the child
* Children with uncomplicated malaria/ fever episodes
* Children whose mothers consent to participate

Exclusion Criteria:

* Children aged less 6 months or greater than 4 years (≥ 5 years)
* Children requiring referral to a health facility (severe malaria, complicated fever episode, convulsions/fits, loss of consciousness, and other danger signs)
* Children whose mothers refuse to consent

Ages: 5 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2000 (Actual)
Dates: Start 2010-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients given prompt effective treatment by CDDs: % of <5-year-old children diagnosed with malaria who receive appropriate ACT treatment within 24 hours of onset of malaria. | 36 months

SECONDARY OUTCOMES:
Coverage of prompt effective treatment: % of <5-year-old children with fever who received ACT treatment within 24 hours of onset of malaria, measured through household surveys. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ndyomugyenyi, MD, Principal Investigator — Ministry of Health, Uganda
Locations (1):
- Rukungiri District, Rukungiri, Rukungiri, Uganda

REFERENCES:
- [Result] Mbonye AK, Ndyomugyenyi R, Turinde A, Magnussen P, Clarke S, Chandler C. The feasibility of introducing rapid diagnostic tests for malaria in drug shops in Uganda. Malar J. 2010 Dec 21;9:367. doi: 10.1186/1475-2875-9-367. PMID 21176131
- [Derived] Lal S, Ndyomugenyi R, Paintain L, Alexander ND, Hansen KS, Magnussen P, Chandramohan D, Clarke SE. Caregivers' compliance with referral advice: evidence from two studies introducing mRDTs into community case management of malaria in Uganda. BMC Health Serv Res. 2018 May 2;18(1):317. doi: 10.1186/s12913-018-3124-8. PMID 29720163